CLINICAL TRIAL: NCT06689774
Title: Using a Pragmatic Randomized Rollout Trial to Evaluate Implementation Strategies to Promote Smoking Treatment and Cancer Prevention for Salvation Army Clients
Brief Title: Salvation Army Tobacco Quit Line Referral Implementation Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-0978; UG3CA293756 (NIH); A534253 (Other: UW- Madison); Protocol Version 11/3/25 (Other: UW- Madison)
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Tobacco Use; Smoking; Smoking Cessation
Keywords: Salvation Army
MeSH Terms: conditions — Tobacco Use; Smoking; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: In this pilot study, both participating Salvation Army sites will receive the experimental enhanced implementation support intervention, with the timing of launch staggered across sites to facilitate refinement of the implementation support intervention. Both sites will start implementing referral to the Wisconsin Tobacco Quit Line without consumer incentives for connecting with the Quit Line immediately, and will add these incentives a few months after launching Quit Line referral. The timing of incentive introduction will be staggered across the 2 pilot sites to permit refinement of the incentive strategy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Wisconsin Tobacco Quit Line (WTQL) Referral Implementation Support (Experimental): Both participating sites in this pilot study will be in this experimental enhanced implementation support arm to help us iteratively enhance the feasibility, acceptability, and sustainability of implementation strategies to support WTQL referral in these sites. Salvation Army personnel at participating sites will receive implementation training and ongoing support to help enhance the fit of WTQL referral in their workflows, culture, and climate, and to enhance staff readiness to connect the consumers they serve with the WTQL. No consumer incentives for connecting with the Quit Line immediately by phone will be offered in this arm so it can serve as active comparator condition for the incentivized arm described below.
  Interventions: Behavioral: Cognitive-Motivational Feedback; Behavioral: Staff Tobacco Quit Line Referral Implementation Support
- Incentivized Immediate Wisconsin Tobacco Quit Line (WTQL) Referral (Experimental): In this experimental condition, Salvation Army personnel will implement an incentive strategy designed to encourage Salvation Army consumers to accept immediate referral to the WTQL. The incentive strategy will be adapted by Salvation Army personnel to fit in the local context, and staff will receive training and ongoing support in implementation of the incentive strategy. The modest incentives will be added in a staggered manner across the 2 Salvation Army sites participating in this pilot trial, after at least 3 months of implementing WTQL referral without consumer incentives for immediate calls.
  Interventions: Behavioral: Cognitive-Motivational Feedback; Behavioral: Staff Tobacco Quit Line Referral Implementation Support; Behavioral: Consumer Incentives for Immediate Referral to a Tobacco Quit Line

INTERVENTIONS:
Behavioral: Cognitive-Motivational Feedback — Salvation Army personnel will be trained to offer adult consumers who use tobacco cognitive-motivational feedback about tobacco use via a no-cost, web-based Qualtrics survey that assesses participant knowledge, beliefs, and priorities and provides feedback to promote knowledge of the costs and risks of smoking and knowledge of the costs and benefits of tobacco use treatment options, including Wisconsin Tobacco Quit Line services. The survey is also designed to help participants weigh the importance of the pros and cons of continuing to use tobacco, and the pros and cons of trying to change their tobacco use.
Behavioral: Staff Tobacco Quit Line Referral Implementation Support — Salvation Army personnel will receive training and will be engaged in efforts to plan, evaluate, adapt, and sustain tobacco treatment referral as part of the social services they provide to adult Salvation Army service consumers who use tobacco. Implementation support will take the form of ongoing engagement of an outreach specialist with a team of Salvation Army personnel and consumers who lead Quit Line referral efforts in the Salvation Army.
Behavioral: Consumer Incentives for Immediate Referral to a Tobacco Quit Line — Salvation Army personnel will offer an incentive to adult consumers who use tobacco to encourage immediate acceptance of a live call with the Wisconsin Tobacco Quit Line. The incentive will be designed by Salvation Army personnel to fit the local context and to be sustainable over time, such as extra access to existing support or resources.
  Arms: Incentivized Immediate Wisconsin Tobacco Quit Line (WTQL) Referral

SUMMARY:
The goal of this clinical trial is to understand how the Salvation Army staff can help people who use tobacco learn about and connect with no-cost treatments to help cut down or quit smoking. Researchers will gather information about the thoughts and experiences of people who smoke tobacco and receive services at the Salvation Army, as well as the experiences of the staff offering support to help treat tobacco use.

DETAILED DESCRIPTION:
In this 2-year pilot study, a team of Salvation Army personnel and consumers will work with a member of the University of Wisconsin Center for Tobacco Research and Intervention Regional Outreach team to plan, implement, and evaluate strategies to connect Salvation Army service consumers with the Wisconsin Tobacco Quit Line for help quitting smoking. The study team will pilot test and refine an enhanced implementation support protocol designed to help Salvation Army teams adapt quitline referral workflows and implementation strategies to fit well with the culture and climate of participating Salvation Army sites, and to enhance Salvation Army staff readiness to connect the consumers they serve with the Wisconsin Tobacco Quit Line. The study team will also pilot test and refine a strategy that Salvation Army personnel can use to incentivize acceptance of Wisconsin Tobacco Quit Line connections by consumers while they are at the Salvation Army service center. To evaluate and enhance the 2 implementation strategies of interest in this study (enhanced implementation support for personnel and an incentive for consumers to accept a connection with the Quit Line while at the Salvation Army), the study team will conduct qualitative interviews with both personnel and consumers at Salvation Army sites, and will collect survey data from personnel and consumers. Service records from both the Salvation Army and Wisconsin Tobacco Quit Line will also be collected for this study to help evaluate the reach of the tobacco treatment intervention, and the representativeness of its reach across subpopulations of consumers. Data regarding the process of implementing Wisconsin Tobacco Quit Line referral in the Salvation Army will also be gathered via observation and recordings of project team meetings. These sources of data will be integrated to help evaluate how well the strategies of interest work in 2 Salvation Army sites, and to refine these in preparation for a full-scale cluster-randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Involved in the management, delivery, or receipt of social services offered by a participating Salvation Army site, or a member of the University of Wisconsin-Center for Tobacco Research and Intervention Outreach Team supporting Wisconsin Tobacco Quit Line implementation
* Able to speak English, Spanish, or another language for which an interpreter is available

Exclusion Criteria:

* Children under the age of 18
* Unable to speak a common language with a study team member or available interpreter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Wisconsin Tobacco Quit Line (WTQL) referral rate | 18 months
  Proportion of adult Salvation Army consumers who use tobacco referred to the WTQL in any modality. Goal is at least 10% without incentives, and at least 16% with incentives.
Wisconsin Tobacco Quit Line (WTQL) enrollment rate | 18 months
  Proportion of clients referred from Salvation Army sites that enroll in WTQL services. Goal is at least 5% without incentives, 8% with incentives.
Salvation Army personnel WTQL referral training engagement | 18 months
  Proportion of eligible Salvation Army personnel who participate in at least some WTQL referral training. Goal is at least 70%.
Tobacco use screening of adult consumers of Salvation Army services | 18 months
  Rate of asking about and documenting current tobacco use among all adult consumers of eligible services in participating Salvation Army sites. Goal is 50% screening rate.

SECONDARY OUTCOMES:
Self-reported abstinence from smoking in the past 7 days | 3 months, 6 months post target date to quit smoking
  Number of WTQL service clients referred from the Salvation Army who report no smoking in the past 7 days at follow-up
Immediate referral via live calls to Wisconsin Tobacco Quit Line (WTQL) | 18 months
  Rate of immediate referral via live calls to WTQL among adult Salvation Army consumers who use tobacco (this will be a subset of the primary referral outcome)
Salvation Army personnel adoption of WTQL referral | 18 months
  Proportion of eligible Salvation Army personnel who refer at least 1 client to the WTQL. Goal is at least 60%.
Cost per successful WTQL referral | 18 months
  Estimated cost of successfully connecting a Salvation Army consumer with the WTQL, with and without incentives for immediate WTQL connection

CONTACTS AND LOCATIONS:
Overall Officials: Danielle McCarthy, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Center for Tobacco Research and Intervention, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual-level original data collected in this trial will be shared. Aggregate data on Salvation Army and Wisconsin Tobacco Quit Line data used in analyses for this trial will also be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: By the time of publication of the primary outcome analyses or the end of the performance period, whichever comes sooner, and up to 7 years after publication.
Access Criteria: IRB approval and meeting restricted use criteria in the data repository.